CLINICAL TRIAL: NCT00503191
Title: Intention-based Therapy for Autism Spectrum Disorder: Promising Results of a Wait-List Control Study in Children
Brief Title: NeuroModulation Technique Treatment of Autism
Acronym: NMT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroModulation Technique Research Institute (Other)
Responsible Party: Principal Investigator, Robert H. Weiner, Ph.D., Principal Investigator, NeuroModulation Technique Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMTRI001-01
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Autism; Neurodevelopmental Disorder
Keywords: Autism; Neurodevelopmental disorder
MeSH Terms: conditions — Autistic Disorder; Neurodevelopmental Disorders

ARMS (1):
- Intention-based therapy treatment for autism (Experimental): NeuroModulation Technique
  Interventions: Behavioral: NeuroModulation Technique

INTERVENTIONS:
Behavioral: NeuroModulation Technique — NeuroModulation Technique is an informational technique that works by identifying and bringing awareness of the mind-body to incorrect informational states of the nervous system which has led to illness or maladaptive behavior. NeuroModulation Technique then directs the body to correct these information states, thereby helping the nervous system resume more adaptive functioning.
  Other Names: NMT

SUMMARY:
The purpose of this study is to determine whether NeuroModulation Technique (NMT) is effective in reducing maladaptive behaviors and increasing adaptive behaviors in children diagnosed with autism.

Hypothesis: Children in the Experimental group will show significant improvement over the Wait-List control group as measured by the Pervasive Developmental Disorder Behavioral Inventory (PDDBI), the Aberrant Behavior Checklist, Community Version (ABC-C), and the Autism Treatment Evaluation Checklist (ATEC). Children in the Wait-List control group will show significant improvement over their baseline measures after receiving NMT treatment.

ELIGIBILITY:
Inclusion Criteria:

* Qualified participants are those who have received a formal diagnosis of autism from a physician or psychologist using DSM-IV, DSM-IV-TR or ICD-9-CM diagnostic criteria. Parents and/or legal guardian must supply proof of autism diagnosis. Autism (DSM-IV, DSM-IV-R or ICD-9-CM 299.0) must be diagnosed - any other diagnosis such as Pervasive Developmental Disorder (PDD), Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS) or Asperger Syndrome is not sufficient for inclusion in this study.
* Children must have had their diagnosis of autism for at least one year prior to the date of the application for participation in this study.
* Children must not have started any new therapies or stopped any ongoing therapies designed to treat their autism such behavior therapy, speech therapy, physical therapy, sensory integration, dietary modification or dietary supplementation, or any alternative or experimental therapies not mentioned here in the 6 months prior to the date of the application for participation in this study.
* During the course of this study, children will be required to continue with any therapies they have been receiving prior to starting the study, and they will be required to not start any new therapies besides NeuroModulation Technique during the course of this study.
* Parents and/or legal guardians of children in the study must be fluent in English and complete all forms and questionnaires in English (for U.S. and Canadian research sites only)

Exclusion Criteria:

* Excluded from participating will be children with any of the following medical conditions: cerebral palsy, Down's syndrome, traumatic brain injury, encephalitis, Lyme disease, cancer, any active infectious disease, endocrine disorder, other mental disorders such as psychotic disorders or other mood disorders including bipolar disorders, or any acute, chronic or unstable medical condition (such as a seizure disorder, Crohn's disease, asthma, bronchitis, etc.) other than autism for which the child has been receiving treatment, medication and/or therapy.
* Also excluded from the study are children who have undergone chelation therapy in the past or are currently undergoing chelation therapy, and children who have displayed significant self-injurious behavior (children who have caused visible harm to themselves).Children with a history of mild to moderate food or airborne allergies, sensitivities, or mild digestive problems are eligible to participate in the study.
* In order to participate in the study, children must not have received any previous NeuroModulation Technique treatment.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2007-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Primary efficacy outcome measures include mean change from start of treatment to end of treatment on the PDDBI Autism Composite Index, the ABC-C Total Score, and the ATEC Total Score. | At the end of 12 NMT treatment sessions.
  Children in both the Experimental and Wait-List control groups will show significant improvement over their respective baseline scores in these primary outcome measures following NMT treatment, which will reflect an improvement in adaptive behaviors as well as a decrease in maladaptive behaviors.

SECONDARY OUTCOMES:
Secondary outcome measures include mean change from start of treatment to end of treatment on the remaining subscales of the PDDBI, the ABC-C, and the ATEC. | At the end of 12 NMT treatment sessions.
  Children in both the Experimental and Wait-List control groups will show significant improvement over their respective baseline scores in these secondary outcome measures following NMT treatment, which will reflect an improvement in adaptive behaviors as well as a decrease in maladaptive behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Weiner, Ph.D., Study Chair — NeuroModulation Technique Research Institute
Locations (1):
- Robert H. Weiner, Ph.D., Dallas, Texas, United States

REFERENCES:
- [Result] Weiner RH, Greene RL. Intention-based therapy for autism spectrum disorder: promising results of a wait-list control study in children. Explore (NY). 2014 Jan-Feb;10(1):13-23. doi: 10.1016/j.explore.2013.10.005. Epub 2013 Oct 17. PMID 24439092
- See also: Study results and parent reports may be found here. — http://www.mind-bodywellnesscenter.org/dr-weiners-autism-research-study/